CLINICAL TRIAL: NCT00096655
Title: A Randomized, Placebo-controlled, Double-blind Trial to Evaluate the Safety and Efficacy of Infliximab in Patients With Active Ulcerative Colitis
Brief Title: A Safety and Efficacy Study for Infliximab (Remicade) in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004783
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Infliximab; Remicade
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of infliximab (Remicade) in patients with Ulcerative Colitis. Infliximab (Remicade) targets specific proteins in the body's immune system to help control the development of inflammation to help reduce painful disease.

DETAILED DESCRIPTION:
This study is designed to investigate the safety and effectiveness of infliximab in adult patients with active ulcerative colitis. The purpose of this study is to see if the symptoms of ulcerative colitis are lessened with this medication infliximab, and what dose is needed to do that safely.Patients will receive infusions of either 5 or 10 mg/kg or placebo at weeks 0, 2, 6, 14, and 22 up to week 164. Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures.

Patients will receive infusions (into the vein) of either 5 or 10 mg/kg or placebo at weeks 0, 2, 6, and every 8 weeks up to week 164.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had ulcerative colitis of at least 3 months' duration at screening, confirmed by the biopsy taken at screening
* Patients must have active colitis confirmed during the screening sigmoidoscopy
* Patients must have active disease.

Exclusion Criteria:

* Patient must not be likely to require surgical removal of all or part of the colon within 12 weeks of beginning the study
* Patient must not require, or required within the 2 months prior to beginning the study, surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intra-abdominal or pancreatic abscess requiring surgical drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2002-05; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with clinical response, defined as a decrease from baseline in the Mayo score by = 30% and = 3 points, with a decrease in the rectal bleeding subscore of = 1 or a rectal bleeding subscore of 0 or 1, at week 8 .

SECONDARY OUTCOMES:
Achievement of clinical remission defined as a Mayo score of = 2 points, with no individual subscore > 1 at week ,Patients in remission will have a rectal bleeding subscore of either 0 or 1, patients who demonstrate mucosal healing at week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Feagan BG, Reinisch W, Rutgeerts P, Sandborn WJ, Yan S, Eisenberg D, Bala M, Johanns J, Olson A, Hanauer SB. The effects of infliximab therapy on health-related quality of life in ulcerative colitis patients. Am J Gastroenterol. 2007 Apr;102(4):794-802. doi: 10.1111/j.1572-0241.2007.01094.x. Epub 2007 Feb 23. PMID 17324131
- [Result] Reinisch W, Sandborn WJ, Bala M, Yan S, Feagan BG, Rutgeerts P, Radford-Smith G, Xu S, Eisenberg D, Olson A, Colombel JF. Response and remission are associated with improved quality of life, employment and disability status, hours worked, and productivity of patients with ulcerative colitis. Inflamm Bowel Dis. 2007 Sep;13(9):1135-40. doi: 10.1002/ibd.20165. PMID 17476675
- [Result] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Derived] Adedokun OJ, Sandborn WJ, Feagan BG, Rutgeerts P, Xu Z, Marano CW, Johanns J, Zhou H, Davis HM, Cornillie F, Reinisch W. Association between serum concentration of infliximab and efficacy in adult patients with ulcerative colitis. Gastroenterology. 2014 Dec;147(6):1296-1307.e5. doi: 10.1053/j.gastro.2014.08.035. Epub 2014 Aug 28. PMID 25173754
- [Derived] Colombel JF, Rutgeerts P, Reinisch W, Esser D, Wang Y, Lang Y, Marano CW, Strauss R, Oddens BJ, Feagan BG, Hanauer SB, Lichtenstein GR, Present D, Sands BE, Sandborn WJ. Early mucosal healing with infliximab is associated with improved long-term clinical outcomes in ulcerative colitis. Gastroenterology. 2011 Oct;141(4):1194-201. doi: 10.1053/j.gastro.2011.06.054. Epub 2011 Jun 30. PMID 21723220
- [Derived] Sandborn WJ, Rutgeerts P, Feagan BG, Reinisch W, Olson A, Johanns J, Lu J, Horgan K, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Colectomy rate comparison after treatment of ulcerative colitis with placebo or infliximab. Gastroenterology. 2009 Oct;137(4):1250-60; quiz 1520. doi: 10.1053/j.gastro.2009.06.061. Epub 2009 Jul 28. PMID 19596014
- See also: A Randomized, Placebo-controlled, Double-blind Trial to Evaluate the Safety and Efficacy of Infliximab in Patients with Active Ulcerative Colitis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=151&filename=CR004783_CSR.pdf
- See also: | A Randomized, Placebo-controlled, Double-blind Trial to Evaluate the Safety and Efficacy of Infliximab in Patients with Active Ulcerative Coliti — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=151&filename=CR004783_REF1.pdf
- See also: A Randomized, Placebo-controlled, Double-blind Trial to Evaluate the Safety and Efficacy of Infliximab in Patients with Active Ulcerative Coliti — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=151&filename=CR004783_REF2.pdf